CLINICAL TRIAL: NCT01401413
Title: A Prospective Randomized, Placebo-Controlled Double-Blind Study to Determine the Efficacy of Ramelteon in REM Sleep Behavior Disorder
Brief Title: Study to Determine Whether Ramelteon Helps People With REM Sleep Behavior Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sleep Medicine Centers of WNY (Other)
Responsible Party: Daniel I Rifkin, MD, President
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEU1640207B
Record Dates: First submitted 2011-07-22; First posted 2011-07-25 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: REM Sleep Behavior Disorder
MeSH Terms: conditions — REM Sleep Behavior Disorder | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): placebo control nightly
  Interventions: Drug: placebo
- 2 (Active Comparator): 8 mg ramelteon nightly
  Interventions: Drug: ramelteon

INTERVENTIONS:
Drug: ramelteon — 8 mg nightly for 30 nights
  Other Names: rozerem
  Arms: 2
Drug: placebo — placebo control i pill nightly for 30 nights
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether the use of the drug ramelteon decreases the symptoms of REM Sleep Behavior Disorder.

DETAILED DESCRIPTION:
This is a randomized double blind placebo controlled study to determine whether the use of ramelteon decreases symptoms of RBD. Outcome measures are determined by change in RBD polysomnographic score and assessment scores on the RBD symptom questionnaire and sleep diary.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for RBD as determined by screening PSG's
* steady bed partner for completion of RBD questionnaire

Exclusion Criteria:

* Hepatic impairment
* RBD associated with narcolepsy
* use of fluvoxamine, rifampin, fluconazole or ketoconazole
* current alcohol or drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change in polysomnographic scores | 30 days

SECONDARY OUTCOMES:
change in RBD symptom questionnaire and sleep diary | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Rifkin, MD, Principal Investigator — Sleep medicine Centers of Western New York
Locations (1):
- Sleep Medicine Centers of WNY, West Seneca, New York, United States